CLINICAL TRIAL: NCT01847911
Title: Self-directed Video Versus Instructor-based Neonatal Resuscitation Training of Novice Providers. A Controlled Blinded Randomized Non-inferiority Multicenter Study
Brief Title: Self-directed Video Versus Instructor-based Neonatal Resuscitation Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Pontifical Catholic University of Argentina (Other); Fisher and Paykel Healthcare (Industry)
Responsible Party: Principal Investigator, Edgardo Szyld, Adjunct Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: GCO 13-1336
Record Dates: First submitted 2013-04-22; First posted 2013-05-07 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2019-01

CONDITIONS: Resuscitation of Newborn Training
Keywords: self instructed resuscitation training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self instructed video learning (Experimental): A complete video lesson of neonatal resuscitation including initial resuscitative maneuvers and administration of ventilation with a SIB and a T-piece resuscitator presented in the primary language of the participating center or university (Spanish or English). A portable kit with a newborn mannequin will be provided for independent video guided practice during the session.
  Interventions: Other: Self instructed video learning
- instructor training (Active Comparator): A standard hands-on training with a face-to-face instructor following a pre-validated OSCE program guidelines.
  Interventions: Other: instructor training

INTERVENTIONS:
Other: Self instructed video learning — A complete video lesson of neonatal resuscitation including initial resuscitative maneuvers and administration of ventilation with a SIB and a T-piece resuscitator presented in the primary language of the participating center or university (Spanish or English). A portable kit with a newborn mannequin will be provided for independent video guided practice during the session.
  Other Names: Self learning video
  Arms: Self instructed video learning
Other: instructor training — a pre-validated OSCE neonatal resuscitation program
  Other Names: face to face training in neonatal CPR
  Arms: instructor training

SUMMARY:
The effect of a self directed video strategy will be compared to a face to face neonatal resuscitation training program. The hypothesis is that both strategies are equivalent.

DETAILED DESCRIPTION:
The NRP is becoming more and more a self learning program followed by a written test and practical hands-on evaluation; but the way the practical skills are taught and practiced has not been uniformly determined.

The current strategies for teaching involve resuscitation instructors. There are several difficulties in the developing world to achieve the objective of having a provider trained in neonatal resuscitation in every delivery. Part of this problem is due to the lack of instructors and-or budget constraint in addition to logistic difficulties.

Our Hypothesis is that a well developed self administered video complemented by a self practice using a mannequin will allow providers to reach at least similar performances on the initial steps and mask ventilation for neonatal resuscitation.

Objectives:

The aim of this study is to test the hypothesis that a self administrated video jointly with a mannequin give similar results than the current Neonatal Resuscitation Program (NRP), a pre-validated Objective Structured Clinical Examination (OSCE)hands-on course provided by a certified instructor.

Specific aim:

To compare the effectiveness of two different teaching strategies on the quality of the ventilation of a mannequin, using a mask by NAÏVE providers. In two different moments, approximately 15 minutes after having taken the course and at a mean of 3 months afterwards.

Two different groups of novice providers will be randomly selected to receive one of the following teaching strategies:

A. A Video based Self instruction with simultaneous video triggered practice with a mannequin without instructor feedback (Spanish in South America, English in North America) on initial steps and adequate mask ventilation for neonatal resuscitation.

B. A pre standardized hands on lesson will be offered by a NRP certified instructor followed by a debriefing session per a pre-validated OSCE protocol (current standard).

Afterwards, all the subjects will be invited to ventilate a mannequin with a standardized instruction (tbd for example…2 minutes ventilation, rate 40 to 60 and the necessary pressure to slightly reach chest rising). This performance will be digitally recorded.

Two independent certified instructors will evaluate the performance, blinded to the assigned group. A previously validated OSCE (objective structured clinical evaluation) performance evaluation grid will be used. The gold standard will consist on a high quality performance done by an NRP instructor.

ELIGIBILITY:
Inclusion Criteria:

* Medical Students from second year and above not previously trained in NRP (the Neonatal Resuscitation Program)
* Nursing Students from second year and above not previously trained in NRP
* Informed consent signed

Exclusion Criteria:

* previous experience in NRP

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2015-11; Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
a pre-validated OSCE | approximately 15 minutes after having taken the course
  proportion of students completing the mandatory fields of the a pre-validated OSCE evaluation grid

SECONDARY OUTCOMES:
a pre-validated OSCE | approximately 15 minutes after having taken the course
  proportion of students approving the OSCE tests
a pre-validated OSCE | at 3 months
  proportion of students approving the OSCE tests
Respiratory rate | approximately 15 minutes after having taken the course
  Respiratory rate provided to the mannequin, number of chest excursions during each performance session.

CONTACTS AND LOCATIONS:
Overall Officials: Egardo G. Szyld, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Demian Szyld, MD, Principal Investigator — New York Simulation Center for the Health Sciences
Locations (7):
- United States (3):
  - New York University Langone Medical Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Oklahoma, Department of Pediatrics, Neonatal-Perinatal Medicine, Oklahoma City, Oklahoma
- Argentina (2):
  - Hospital Universitario Austral, Pilar, Buenos Aires
  - Hospital Italiano, Buenos Aires, City of Buenos Aires
- Pontificia Universidad Catolica de Chile, Santiago, Chile
- Universidad de las Americas Puebla, San Andrés, Cholula, Mexico

REFERENCES:
- [Result] Szyld EG, Aguilar A, Lloret SP, Pardo A, Fabres J, Castro A, Dannaway D, Desai PV, Capelli C, Song CH, Enriquez D, Szyld D; EdM on behalf of the SAVER Study Group. Self-directed video versus instructor-based neonatal resuscitation training: a randomized controlled blinded non-inferiority multicenter international study. J Perinatol. 2021 Jul;41(7):1583-1589. doi: 10.1038/s41372-021-00941-x. Epub 2021 Feb 15. PMID 33589725